CLINICAL TRIAL: NCT02362295
Title: Prospective National Survey of the Palliative Situation Among Inmates in French Prisons
Acronym: PARME
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Hospices Civils de Lyon (Other); Central Hospital, Nancy, France (Other); University Hospital, Lille (Other); University Hospital, Marseille (Other); University Hospital, Toulouse (Other); University Hospital, Bordeaux (Other); Rennes University Hospital (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Régis AUBRY, professor, Centre Hospitalier Universitaire de Besancon
Other Study IDs: 2011-A00791-40
Record Dates: First submitted 2015-02-09; First posted 2015-02-12 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Critical Illness; Terminal Illness
Keywords: palliative care; vulnerable population; qualitative research
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- census: qualitative interview
  Interventions: Other: qualitative interview

INTERVENTIONS:
Other: qualitative interview — some patient are interviewed.

SUMMARY:
PARME study had 3 objectives:

* To identify the specific number of incarcerated individuals with terminal illness in need of palliative care.
* To describe the health and penal situation of these prisoners.
* To analyse the situation of these ill prisoners especially in the context of suspended sentence for medical ground

In order to answer these questions, the investigators used a mixed method research.

DETAILED DESCRIPTION:
First, in order to establish a baseline, the investigators contacted the medical units in all French prisons, which means 178 care units and 8 secures inpatient care units. The investigators census every patient with terminal illness, which was defined in this study as an evolutive pathology with a life prognosis less than a year.

A questionnaire was completed by these physicians for every situation. The census was conducted for three months across France.

For the qualitative study, the investigators selected 14 specific situations chosen into these which had been identified by the physicians.

The investigators wanted to get 3 types of patients :

1. patient who had obtained a compassionate release
2. patient whose demand has been refused
3. patient who did not demand any release. The four interviews (patients, physisians, judges, probation workers) for each situation has explained the global situation.

Each interviewee spoke about the situation with his/her perspective and sense that they attributed to the actions of others.

This research analyzes the particularity of each of these end of life situations in prison.

ELIGIBILITY:
Inclusion Criteria:

* prisonners
* serious and evolving pathology
* vital prognosis less than a year

Exclusion Criteria:

* less than 18 year
* person under tutelage
* patient who refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every prisonners with terminal illness
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-05; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
census ill prisonners with vital prognosis less than a year and understand how penal and medical professional are coping with these situations | 1 year

SECONDARY OUTCOMES:
uderstand how professionnels are coping with not condamned prisonners | 1 year
Question the meaning of the sentence for ill prisonners | 1 year
Compare the way professionnal are coping with these situation around France | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Amzallag, Dr, Principal Investigator — Hospices Civils de Lyon; Sebastien Grignard, Dr, Principal Investigator — Centre Hospitalier Universitaire de Besancon; Blanchet Emmanuelle, Dr, Principal Investigator — CHU NANCY; Grimopont Frederic, Dr, Principal Investigator — CHU Lille; Bartoli Christophe, Dr, Principal Investigator — CHU Marseille; BAYLE Paule, Dr, Principal Investigator — University Hospital, Toulouse; Bedry Regis, Dr, Principal Investigator — University Hospital, Bordeaux; Bernard Benoit, Dr, Principal Investigator — CHU Rennes; Auger Yvain, Dr, Principal Investigator — APHP

REFERENCES:
- [Background] AUBRY R., 2011, Etat des lieux du développement des soins palliatifs en France en 2010, Rapport à M. Le Président de la République, M. Le Premier Ministre, Comité national de suivi du développement des soins palliatifs.
- [Background] BERTRAND D, NIVEAU G, 2006, Santé et Prison. Chêne-Bourg : Editions Médecine & Hygiène, 2006
- [Background] Bolger M. Dying in prison: providing palliative care in challenging environments. Int J Palliat Nurs. 2005 Dec;11(12):619-20; discussion 621. doi: 10.12968/ijpn.2005.11.12.20227. PMID 16415753
- [Background] Byock I. Dying well in corrections: why should we care? Correctcare. 2002 Fall;16(4):18. No abstract available. PMID 12705265
- [Background] Chow RK. Initiating a long-term care nursing service for aging inmates. Geriatr Nurs. 2002 Jan-Feb;23(1):24-7. doi: 10.1067/mgn.2002.122562. PMID 11865254
- [Background] Cohn F. The ethics of end-of-life care for prison inmates. J Law Med Ethics. 1999 Fall;27(3):252-9, 210. doi: 10.1111/j.1748-720x.1999.tb01459.x. PMID 11067602
- [Background] DARBEDA P., mars-juin 1999, " Médecine et détenus ", Journal international de bioéthique, n°1-2, pp 35-45.
- [Background] Drescher GP. Prisoner's right to refuse treatment outweighs physician's duty to treat. J Law Med Ethics. 1993 Fall-Winter;21(3-4):400-1. No abstract available. PMID 11654964
- [Background] Dubler NN. The collision of confinement and care: end-of-life care in prisons and jails. J Law Med Ethics. 1998 Summer;26(2):149-56. doi: 10.1111/j.1748-720x.1998.tb01670.x. No abstract available. PMID 11657351
- [Background] Finlay IG. Managing terminally ill prisoners: reflection and action. Palliat Med. 1998 Nov;12(6):457-61. doi: 10.1191/026921698674823377. PMID 10621866
- [Background] Gallagher EM. Elders in prison. Health and well-being of older inmates. Int J Law Psychiatry. 2001 Mar-Jun;24(2-3):325-33. doi: 10.1016/s0160-2527(00)00080-7. No abstract available. PMID 11436633
- [Background] Kiel RA. Caring for terminally ill inmates: on-site hospice care or compassionate release? Correctcare. 1995 Jun-Jul;9(2):5, 13-14. No abstract available. PMID 11660066
- [Background] Lin J, Mathew P. Prison inmates and palliative care. JAMA. 2007 Dec 5;298(21):2481; author reply 2481. doi: 10.1001/jama.298.21.2481-a. No abstract available. PMID 18056900
- [Background] Lincoln A. Improving the conditions of confinement. End-of-life care in prison. Pharos Alpha Omega Alpha Honor Med Soc. 2008 Autumn;71(4):18-25. No abstract available. PMID 19014115
- [Background] Linder JF, Meyers FJ. Palliative care for prison inmates: "don't let me die in prison". JAMA. 2007 Aug 22;298(8):894-901. doi: 10.1001/jama.298.8.894. PMID 17712073
- [Background] Lum KL. Palliative care behind bars: the New Zealand prison hospice experience. J Pain Palliat Care Pharmacother. 2003;17(3-4):131-8; discussion 139-40. PMID 15022957
- [Background] Mahon NB. Introduction: death and dying behind bars--cross-cutting themes and policy imperatives. J Law Med Ethics. 1999 Fall;27(3):213-5. doi: 10.1111/j.1748-720x.1999.tb01454.x. No abstract available. PMID 11067597
- [Background] Mara CM. Expansion of long-term care in the prison system: an aging inmate population poses policy and programmatic questions. J Aging Soc Policy. 2002;14(2):43-61. doi: 10.1300/J031v14n02_03. PMID 12557993
- [Background] MOUQUET M-C, 2005 (mars), " La santé des personnes entrées en prison en 2003 ",Études et résultats, n°386, DREES.
- [Background] MOUQUET M-C, DUMONT M., BONNEVIE M-C, 1999 (janvier)" La santé à l'entrée en prison, un cumul des facteurs de risques ", Études et résultats, n°4, DREES.
- [Background] O'Connor MF. Finding boundaries inside prison walls: case study of a terminally ill inmate. Death Stud. 2004 Jan;28(1):63-76. doi: 10.1080/07481180490249274. PMID 14969279
- [Background] Ratcliff M, Craig E. The GRACE Project: Guiding End-of-Life Care in Corrections 1998-2001. J Palliat Med. 2004 Apr;7(2):373-9. doi: 10.1089/109662104773709549. PMID 15130219
- [Background] SANDO ROY (de) B., 2004 (mars), " La suspension de peine pour raison médicale : Une parenthèse de la peine contre une parenthèse de la santé. ", Droit Déontologie & Soin.; 4(1), pp 4-15.
- [Background] Reeder D, Meldman L. Conceptualizing psychosocial nursing in the jail setting. J Psychosoc Nurs Ment Health Serv. 1991 Aug;29(8):40-4. doi: 10.3928/0279-3695-19910801-10. PMID 1920202
- [Background] SANNIER O, MANALOUIL C., 2008, " Est-ce que le secret médical est la clé de voûte du respect de l'éthique médicale en prison ? ", Éthique & Santé; 5(4), pp201-207.
- [Background] Snow T. Should dying prisoners be given their freedom for a more dignified end? Nurs Stand. 2009 Aug 26-Sep 1;23(51):12-3. No abstract available. PMID 19753771
- [Background] TRAULLE É, WERBROUCK A, MANAOUIL C., 2006 (sept) " La suspension de peine pour raison médicale. " Médecine & Droit., 79-80, pp 142-146.
- [Background] Turner M, Barbarachild Z, Kidd H, Payne S. How notorious do dying prisoners need to be to receive high quality end-of-life care? Int J Palliat Nurs. 2009 Oct;15(10):472-3. doi: 10.12968/ijpn.2009.15.10.44884. No abstract available. PMID 20081718
- [Background] Vesely R. Another aging population. More states considering early-release programs for older, infirm inmates. Mod Healthc. 2010 Mar 29;40(13):32-3. No abstract available. PMID 20380057
- [Background] Zelaya E. The challenges of caring for an incarcerated patient. Am J Hosp Palliat Care. 2009 Jun-Jul;26(3):230-1. doi: 10.1177/1049909109333931. No abstract available. PMID 19531700
- [Background] Wilford T. Developing effective palliative care within a prison setting. Int J Palliat Nurs. 2001 Nov;7(11):528-30. doi: 10.12968/ijpn.2001.7.11.9292. PMID 11775927
- [Background] Wood FJ. The challenge of providing palliative care to terminally ill prison inmates in the UK. Int J Palliat Nurs. 2007 Mar;13(3):131-5. doi: 10.12968/ijpn.2007.13.3.23275. PMID 17505406
- [Background] ZIMMERAMANN N., WALD F.S., THOMPSON A.S., 2002 (juillet), " The needs and ressources for hospice care in the connecticut prison system : a feasibility study. ", Illness, Crisis and Cross, vol 10, n°3, pp204-232.
- [Derived] Rothman A, McConville S, Hsia R, Metzger L, Ahalt C, Williams BA. Differences between incarcerated and non-incarcerated patients who die in community hospitals highlight the need for palliative care services for seriously ill prisoners in correctional facilities and in community hospitals: A cross-sectional study. Palliat Med. 2018 Jan;32(1):17-22. doi: 10.1177/0269216317731547. Epub 2017 Sep 27. PMID 28952889
- [Derived] Pazart L, Godard-Marceau A, Chassagne A, Vivot-Pugin A, Cretin E, Amzallag E, Aubry R; PARME Study Group. Prevalence and characteristics of prisoners requiring end-of-life care: A prospective national survey. Palliat Med. 2018 Jan;32(1):6-16. doi: 10.1177/0269216317721816. Epub 2017 Aug 8. PMID 28786339